CLINICAL TRIAL: NCT01653938
Title: A Randomized Controlled Trial of a CPR Video in Heart Failure Patients
Brief Title: A Trial of a CPR Video in Heart Failure Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-P-002083
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention)
- Video Arm (Experimental): Use of video decision aid in the experimental arm.
  Interventions: Behavioral: video decision aid

INTERVENTIONS:
Behavioral: video decision aid
  Arms: Video Arm

SUMMARY:
This is a randomized controlled trial of a CPR video decision aid in patients with advanced congestive heart failure (CHF).

DETAILED DESCRIPTION:
Aim 1: To compare the care preferences for CPR and intubation among subjects randomized to video and subjects randomized to the current standard of care without the video.

Hypothesis 1: Subjects randomized to the video intervention will be significantly more likely to opt against CPR and intubation compared to those who do not see the video.

Aim 2: To compare code-status documentation in the electronic medical records between subjects randomized to the video and those who are receiving the current standard of care without the video.

Hypothesis 2: Subjects randomized to the video are more likely to have their code status correctly documented in the electronic medical records compared to those who do not see the video.

Aim 3: To compare knowledge and decisional conflict of subjects randomized to video and subjects randomized to the current standard of care without the video.

Hypothesis 3: When compared to subjects randomized to the current standard of care, subjects in the video intervention group will have higher knowledge and lower decisional conflict (lower decisional conflict scores) when asked to choose CPR and intubation preferences.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of advanced heart failure:

   * New York Heart Association Class III or IV (III: marked limitation in activity due to symptoms, even during less-than-ordinary activity; IV: severe limitations, experiences symptoms while at rest). AND
   * Two or more hospitalizations for heart failure in the last year. AND
   * Either a systolic blood pressure ≤ 120 mm Hg OR Na ≤ 135 mEq/L.
2. Ability to provide informed consent.
3. Ability to communicate in English.
4. Age 65 or older.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
preferences | 5 minutes after survey
  preferences for cpr and intubation

SECONDARY OUTCOMES:
knowledge | 5 minutes after survey
  knowledge of cpr and intubation
decisional conflict | 5 minutes after survey
  decisional conflict
advance care planning documentation | by the end of one year
  advance care planning in medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States